CLINICAL TRIAL: NCT04857580
Title: Intracoronary Cryotherapy Effect for staBilization of vulnErable Plaque at Risk of Rupture as Assessed by imaGing
Brief Title: Pilot Study on the Effect of Intracoronary Cryotherapy on Stabilization of Vulnerable Plaque at Risk of Rupture
Acronym: ICEBERG
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: Cryotherapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-CD-P01-1
Record Dates: First submitted 2021-04-13; First posted 2021-04-23 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTS device (Experimental)
  Interventions: Device: CTS Device
- Control (No Intervention)

INTERVENTIONS:
Device: CTS Device — Coronary cryotherapy is delivered locally on eligible lesions randomized to the treatment using the CTS System.
  Arms: CTS device

SUMMARY:
Atherosclerosis is a progressive inflammatory disease of the large and medium sized arteries, which is characterized by the formation of plaques in the vessel wall. The morphology and composition of the plaque play a major role in its stability during the development of the disease.

The CTS system allows to deliver coronary cryotherapy intended for stabilization of vulnerable plaque with non-significant stenosis. Vulnerable plaque at high risk of rupture will be assessed by NIRS-IVUS imaging modality in patients with Acute Coronary Syndrome (ACS).

The ICEBERG study is an early feasibility single arm study enrolling a maximum of 45 patients. After enrolment of the first 5 patients in the First-in-Man safety cohort, the trial will enroll and randomize 40 eligible lesions in the randomized cohort of which 20 will be treated with cryotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years old.
* Acute cardiac pain/angina consistent with acute coronary syndrome eligible for coronary angiography meeting one of the following criteria:

  1. Non ST-segment elevation myocardial infarction (NSTEMI) with rise/fall of cardiac enzymes (troponin I or T) with at least one value above the 99th percentile of the upper reference limit requiring Percutaneous Coronary Intervention (PCI) within 72 hours from diagnosis
  2. Stabilized ST-segment elevation myocardial infarction (STEMI) with at least one value above the 99th percentile of the upper reference limit requiring PCI within < 12 hours from symptoms onset.
  3. Unstable angina with new or worsening angina symptoms over the last 2 weeks requiring PCI within 72 hours.
* Patient must have one, two or three-vessel disease in native coronary arteries.
* PCI of the culprit lesion on all patients.
* At least one lesion meeting the criteria below:

  1. Located in a non-culprit vessel, or proximal to the culprit lesion if located in the culprit vessel with at least 10 mm distance from the culprit lesion.
  2. Lesion stenosis ≤ 70% of the reference vessel diameter by visual assessment on coronary angiogram.
  3. Plaque-level maxLCBI4mm ≥ 325 by NIRS (Near-Infrared Spectroscopy).
  4. Plaque burden ≥ 65% by IVUS (IntraVascular UltraSound).
  5. Not intended for revascularization based on angiographic criteria and negative physiology assessment (FFR>0.80 or iFR/RFR>0.89).
  6. Lesion-level balloon to artery ratio > 1.0.
  7. Lesion length ≤ 20 mm.
  8. Investigator considers that lesions are accessible.
  9. If more than two suitable lesions available, investigator will select two lesions for randomization.
* Subject able to consent and has a signed and dated the informed consent form.

Exclusion Criteria:

* Unstable patients (cardiogenic shock, hypotension needing inotropes, hypoxia needing intubation, refractory ventricular arrhythmias, and IABP).
* Patients with ongoing ST-segment elevation myocardial infarction.
* Patients that had a procedural complication during the PCI procedure, such as coronary dissection, perforation or a complication that would necessitate immediate and/or unplanned surgical revascularization.
* History of Coronary Artery Bypass Graft (CABG) or planned CABG within 12 months after the index procedure.
* Known ejection fraction < 30%.
* Known severe valvular heart disease.
* Known severe renal insufficiency (eGFR <30 ml/min/1.72 m2).
* Any life-threatening conditions or medical comorbidity resulting in life expectancy < 12 months.
* Participation in any investigational study that has not yet reached its primary endpoint.
* Women who are pregnant or lactating, or NOT surgically sterile (tubal ligation or hysterectomy) or NOT postmenopausal for at least 6 months or women with childbearing potential without effective contraception (pill, patch, ring, diaphragm, implant and intrauterine device).

Angiographic exclusion criteria:

* Visible distal embolization/no-reflow following culprit PCI.
* Left main coronary artery disease (visual diameter stenosis > 50%).
* Stent thrombosis/restenosis as a culprit lesion.
* Index lesion involving a bifurcation.
* Angiographic evidence of severe calcification and/or marked tortuosity of the index vessel and/or lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Cryotherapy procedure related complication | 90 days
  Any cryotherapy procedure related complication defined as coronary artery dissection, acute vessel closure, ischemia, arrythmia, need for bailout stenting, or any Major Adverse Cardiac Events (MACE) adjudicated to the index lesion
Optical Coherence Tomography (OCT)-assessed fibrous cap thickness | 90 days
  Change in Optical Coherence Tomography (OCT)-assessed fibrous cap thickness from index lesion.

SECONDARY OUTCOMES:
Cryotherapy related complication | 9 months
  Any cryotherapy related complication defined as coronary artery dissection, acute vessel closure, ischemia, arrythmia, need for bailout stenting, or any MACE defined as cardiac death, myocardial infarction, revascularization, rehospitalization for unstable or progressive angina adjudicated to the index lesion.
Device success | Baseline
  Device success defined as ability to successfully track and treat the lesion.
Cryotherapy/lesion procedure success | Baseline
  Cryotherapy/lesion procedure success defined as TIMI 3 flow, percent diameter stenosis equivalent to or lower than pre-procedure.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Zealand University Hospital, Roskilde
- Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erlinge D, Maehara A, Ben-Yehuda O, Botker HE, Maeng M, Kjoller-Hansen L, Engstrom T, Matsumura M, Crowley A, Dressler O, Mintz GS, Frobert O, Persson J, Wiseth R, Larsen AI, Okkels Jensen L, Nordrehaug JE, Bleie O, Omerovic E, Held C, James SK, Ali ZA, Muller JE, Stone GW; PROSPECT II Investigators. Identification of vulnerable plaques and patients by intracoronary near-infrared spectroscopy and ultrasound (PROSPECT II): a prospective natural history study. Lancet. 2021 Mar 13;397(10278):985-995. doi: 10.1016/S0140-6736(21)00249-X. PMID 33714389
- [Background] Stone GW, Maehara A, Ali ZA, Held C, Matsumura M, Kjoller-Hansen L, Botker HE, Maeng M, Engstrom T, Wiseth R, Persson J, Trovik T, Jensen U, James SK, Mintz GS, Dressler O, Crowley A, Ben-Yehuda O, Erlinge D; PROSPECT ABSORB Investigators. Percutaneous Coronary Intervention for Vulnerable Coronary Atherosclerotic Plaque. J Am Coll Cardiol. 2020 Nov 17;76(20):2289-2301. doi: 10.1016/j.jacc.2020.09.547. Epub 2020 Oct 15. PMID 33069847